CLINICAL TRIAL: NCT06359821
Title: A Study to Evaluate Safety, Whole-Body Distribution and Radiation Dosimetry of ZA-001, an Alpha-particle-emitting (At211) Radiopharmaceutical, in Metastatic Castration Resistant Prostate Cancer
Brief Title: Evaluate Safety, Whole-Body Distribution and Radiation Dosimetry in Metastatic Castration Resistant Prostate Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Rong Tian, MD, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Z-001
Record Dates: First submitted 2024-04-07; First posted 2024-04-11 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Prostate Cancer
Keywords: PSMA positive metastatic prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single dose (Experimental): ZA-001, single dose
  Interventions: Drug: ZA-001

INTERVENTIONS:
Drug: ZA-001 — Study drug ZA-001 administered via intravenous injection.

SUMMARY:
A Study to Evaluate Safety, Whole-Body Distribution and Radiation Dosimetry of ZA-001, an Alpha-particle-emitting (At211) Radiopharmaceutical, in metastatic castration resistant prostate cancer

ELIGIBILITY:
Inclusion Criteria:

1. Participants provide signed informed consent and confirm that they are able and willing to comply with all protocol requirements.
2. Participants must be ≥18 years of age and competent to give informed consent.
3. Participants must have progressive mCRPC with histologically or cytologically confirmed adenocarcinoma of the prostate. Participants must have documented PSA and/or radiographic progression.
4. Participants must have Gallium 68 PSMA-11 (Ga 68 PSMA-11) Positron Emission Tomography (PET)/Computed Tomography (CT) prostate-specific membrane antigen (PSMA) positive lesions ≤ 30 days prior to beginning study therapy.
5. Participant has not received any form of prostate-cancer directed therapy since undergoing screening PSMA scan.
6. Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
7. Participants must have a life expectancy of more than 3 months.
8. Effective castration with testosterone level of <50 ng/dL and plan to continue with chronic medical or surgical castration.
9. Participants must have adequate hematological and organ function.

Exclusion Criteria:

1. Participants with any medical condition or other circumstances that, in the opinion of the investigator, would preclude participation in this study, compromise obtaining reliable data, achieving study objectives, or completion.
2. Pathological findings consistent with small cell and/or neuroendocrine carcinoma of the prostate or any other histology not consistent with prostate adenocarcinoma.
3. Participants with any PSMA-negative metastatic lesion these criteria were ineligible.
4. Less than 4 weeks since last myelosuppressive therapy (including prior radiotherapy or prior treatment with 223Radium, 89Strontium or 153Samarium containing compounds).
5. With active or uncontrolled infection.
6. Have used any other investigational drugs within 4 weeks or 5 half-lives (whichever is shorter) prior to the start of the study treatment, or have used any investigational medical devices within 4 weeks prior to the start of the study treatment, and plan to receive other investigational drugs or medical devices during the course of this study.
7. Previously known to have a history of allergy, hypersensitivity, or intolerance to radioactive drugs; or known to be allergic to ethanol.
8. Participants who have a pregnant partner or are capable of fathering a child and who are unwilling to take precautions to prevent potential harm to the fetus or prevent pregnancy during and for 90 days after discontinuation of study treatment.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2024-05-17 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2024-10-14 (Actual)

PRIMARY OUTCOMES:
The absorbed radiation doses (Gray [Gy] /Megabecquerel [MBq] )for whole body and organ | 24 hours
  SPECT/CT will be scanned following administration of the ZA-001
Adverse Event | 1 week
  Number of participants with Adverse Events as a measure of safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Rong Tian, MD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Chengdu, China

IPD SHARING:
Plan to Share IPD: No